CLINICAL TRIAL: NCT06403969
Title: SLEEP - in Children With Autism and Intellectual Disability: Investigation and Treatment
Brief Title: Sleep in Children With Autism and Intellectual Disability
Acronym: SLEEP-AID IT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Värmland County Council, Sweden (Other Government)
Collaborators: Uppsala University (Other); Uppsala County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 281174
Record Dates: First submitted 2024-04-10; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Insomnia; Autism; Intellectual Disability
Keywords: applied behavior analysis; polysomnography; insomnia; autism
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Autistic Disorder; Intellectual Disability | interventions — Applied Behavior Analysis

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single case experimental arm (Experimental): ABA intervention with multiple baselines and follow up measurements
  Interventions: Behavioral: Applied Behavior Analysis

INTERVENTIONS:
Behavioral: Applied Behavior Analysis — Applied Behavior Analysis focusing on nocturnal awakenings. It starts with identification of target behaviors and goals. A functional analysis is conducted to analyze the underlying function of a behavior in connection to the problem. A treatment plan is formulated, including strategies to achieve the goals, and methods to evaluate. Families receive education sleep hygiene. Adaptations focus on antecedents and consequences, with an emphasis on positive reinforcement of favorable behaviors. Various components of Cognitive Behavioral Therapy may be applicable. These include changes in sleep environment, stimulus control, bedtime routines with visual support and prompting. Sleep restriction and bedtime fading are included. Modified extinction techniques with parental presence can be applied, gradually phasing out parental immediate presence. The intervention continues until goals are achieved or for a maximum of 8 sessions (each lasting up to 60 minutes) spread over 8 weeks.

SUMMARY:
Purposes: Establish proof-of-concept for home polysomnography in the assessment of sleep disorders among prepubertal school children with autism and intellectual disabilities combined; To explore the diagnostic yield of polysomnography for these individuals; To examine the feasibility and treatment effect of Applied Behavior Analysis (ABA) for insomnia, focusing on sleep maintenance difficulties, in these children.

Method: Single-case experimental design with multiple baselines and with multiple participants, with a focus on feasibility. N=15 prepubertal children, aged 6-12 years, with autism and intellectual disabilities combined, and difficulties in maintaining nighttime sleep. Assessment with home polysomnography + actigraphy. Intervention with ABA, including functional analysis, measurable goals, and behavior modification based on the functional analysis. Outcome measures from actigraphy and sleep diary with multiple data points at baseline and after treatment. Feasibility is examined as adherence to assessment and treatment, as well as in a qualitative study of parental experiences.

DETAILED DESCRIPTION:
Pilot study with a feasibility focus using a single-case experimental design, employing multiple baselines and involving multiple participants. Children aged 6-12 with autism and intellectual disabilities, along with sleep maintenance difficulties, are recruited. Following diagnostic assessment of insomnia, up to two weeks of sleep registration using sleep diaries and actigraphy is initiated. Polysomnography will be used to identify, characterize, and map out the sleep disorder. Registration is conducted at home over one night and supplemented with a home visit. If no significant physiological explanations are discovered, treatment with Applied Behavior Analysis (ABA) conducted by a psychologist is then commenced. The intervention begins with goal formulation. Subsequently, a functional analysis is carried out to analyze the underlying function of a behavior contributing to and maintaining the sleep disorder. This assessment follows the ABC model and is based on clinical interviews, observations, sleep diaries, and actigraphy. Next, a treatment plan with measurable goals and strategies to achieve them is formulated. Interventions are based on both antecedents and consequences, with a strong emphasis on positive reinforcement of favorable sleep behaviors. Overall, the intervention is individualized, and most treatment components from cognitive behavioral therapy may be relevant. Examples include education in sleep hygiene, changes in the sleep environment, and positive reinforcement of favorable behaviors. Stimulus control techniques, such as going to bed when tired and establishing good bedtime routines with visual support, are included. Sleep restriction, limiting naps, and bedtime fading are also part of the intervention. Modified extinction techniques with parental presence may be applied, especially if co-sleeping is problematic, gradually phasing out immediate parental presence in or near the bed while remaining responsive to the child's need for security, with a clear intention to cease co-sleeping. The intervention continues until treatment goals are achieved or for a maximum of eight sessions (up to 60 minutes each) spread over a maximum of eight weeks. Sleep diaries are continued daily throughout the study period, including up to two weeks after the intervention ends. Actigraphy registration is restarted one week after the intervention ends and continues for the same duration as during the baseline registration. Sleep diaries are also recorded in the same manner for a follow-up three months after the intervention ends.

Primary outcomes are change from baseline to follow up one week after completed intervention, regarding Total Sleep Time (TST), Wakefulness After Sleep Onset (WASO), and frequency of night-time awakenings, based on actigraphy. Secondary outcomes are change from baseline to follow up regarding TST, WASO, night-time awakenings and sleep efficiency, based on sleep diaries. Specified outcome is also feasibility of investigation and intervention, as below.

Feasibility of the sleep assessment, including polysomnography, is evaluated in terms of frequency and proportion of completed assessments, as well as parental acceptance of the assessment in the qualitative component below. Method adaptation needs are described. The diagnostic yield of the assessment is reported, patient by patient, and summarized with a hypothesis-generating approach. Parents' experiences of the intervention and its feasibility are qualitatively explored and described. The interview is semi-structured, conducted one month after the intervention ends, and analyzed using qualitative content analysis. Feasibility of the ABA intervention is also evaluated in terms of frequency of completed treatments, therapist ratings of families' adherence to treatment, intervention duration, and therapists' adherence to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Insomnia AND
* Autism AND
* Intellectual Disability.

Exclusion Criteria:

* Started puberty OR
* Epilepsy OR
* Ongoing melatonin treatment OR
* Obstructive sleep apnea

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2024-05-14 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Total Sleep Time | One week after completed intervention,
  Change from baseline to follow up regarding Total Sleep Time (TST), based on actigraphy.
Wakefulness After Sleep Onset | One week after completed intervention,
  Change from baseline to follow up regarding Wakefulness After Sleep Onset (WASO) based on actigraphy
Night time awakenings | One week after completed intervention,
  Change from baseline to follow up regarding Night time awakenings based on actigraphy

SECONDARY OUTCOMES:
Sleep diary measures of Total Sleep Time | One week after completed intervention
  Change from baseline to follow up regarding Total Sleep Time (TST), based on sleep diaries.
Sleep diary measures of Wakefulness After Sleep Onset | One week after completed intervention
  Change from baseline to follow up regarding Wakefulness After Sleep Onset (WASO) based on sleep diary
Sleep diary measures of Night time awakenings | One week after completed intervention
  Change from baseline to follow up regarding nighttime awakenings based on sleep diary

CONTACTS AND LOCATIONS:
Overall Officials: Sverre Wikström, Principal Investigator — Region Värmland

IPD SHARING:
Plan to Share IPD: No